CLINICAL TRIAL: NCT04583111
Title: The Effect of Antiemetics on Bowel Preparation Before Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, Deputy director of the Division of Gastroenterology and Hepatology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RJYYXHNK-006
Record Dates: First submitted 2020-09-22; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Domperidone; Sulpiride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Domperidone group (Experimental): Patients in Domperidone group took 10mg of domperidone 30min before PEG.
  Interventions: Drug: Domperidone
- Sulpiride group (Experimental): Patients in Sulpiride group took 100mg of sulpiride 30min before PEG.
  Interventions: Drug: sulpiride
- Control group (No Intervention): Patients in Control group followed the regular routine of 3L split-dose of PEG.

INTERVENTIONS:
Drug: Domperidone — Domperidone and sulpiride are antiemetics that may be useful in preventing the PEG-related nausea and vomiting.
  Arms: Domperidone group
Drug: sulpiride — Domperidone and sulpiride are antiemetics that may be useful in preventing the PEG-related nausea and vomiting.
  Arms: Sulpiride group

SUMMARY:
Polyethylene glycol (PEG) is one of the most common laxatives used in colonoscopy. However, 5 - 15% of patients can not complete the preparation due to its poor taste and large volume. So this study is aimed to explore the effect of antiemetics on abdominal discomforts associated with PEG.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years patients scheduled for colonoscopy

Exclusion Criteria:

* intestinal obstruction or hemorrhage;
* allergy to domperidone, sulpiride or PEG;
* pregnancy or breastfeeding;
* previous use of prokinetics within 1 month.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the discomforts during bowel preparation | before colonoscopy
  The primary endpoint of this study was the discomforts during bowel preparation such as nausea, vomit, abdominal fullness and pain. These symptoms were assessed as none, mild, moderate and severe. Patients with mild to severe symptoms were classified as presence of discomforts.

SECONDARY OUTCOMES:
The quality of bowel preparation assessed by Boston Bowel Preparation Scale | during colonoscopy
  The secondary endpoint was the quality of bowel preparation assessed by the Boston Bowel Preparation Scale (BBPS) during the withdrawal phase of colonoscopy. The BBPS uses a 0-3 points scale assessing the bowel preparation quality in 3 segments of the colon (the right, transverse and left colons). BBPS score ≥ 6 were defined as adequate bowel preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengliang Chen, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided